CLINICAL TRIAL: NCT02428257
Title: Hypobaric Rather Than Isobaric Bupivacaine to Prevent Anesthesia-induced Hypotension in Patients Undergoing Surgical Repair of Hip Fracture Under Continuous Spinal Anesthesia: a Prospective Randomized Controlled Study.
Brief Title: Continuous Spinal Anesthesia With Hypobaric Bupivacaine to Preserve Hemodynamics in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Kassab d'Orthopédie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P-2015008AR
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Hip Fracture; Hypotension
Keywords: hip fracture; elderly; continous spinal anesthesia; hypobaric bupivacaine; isobaric bupivacaine; hypotension
MeSH Terms: conditions — Hip Fractures; Hypotension | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- hypobaric (Experimental): continuous spinal anesthesia with 2,5 mg boluses of hypobaric bupivacaine, prepared diluting each 1 ml of 0.5% isobaric bupivacaine with 1 ml of sterile water.
  Interventions: Procedure: continuous spinal anesthesia; Drug: hypobaric bupivacaine; Drug: ephedrine
- isobaric (Active Comparator): continuous spinal anesthesia with 2,5 mg boluses of 0.5% isboaric bupivacaine
  Interventions: Procedure: continuous spinal anesthesia; Drug: isobaric bupivacaine; Drug: ephedrine

INTERVENTIONS:
Procedure: continuous spinal anesthesia — Spinal puncture performed with a 19-gauge Tuohy needle at the L4-L5 or L3-L4 interspace using a midline approach. 3 cm of a 22-gauge catheter introduced through the needle, directed to the fractured side.
Drug: hypobaric bupivacaine — hypobaric bupivacaine was prepared diluting each 1 ml of 0.5% isobaric bupivacaine with 1 ml of sterile water.
  Arms: hypobaric
Drug: isobaric bupivacaine — 0.5% isobaric bupivacaine
  Arms: isobaric
Drug: ephedrine

SUMMARY:
The study evaluates the potential beneficial effects on hemodynamics when hypobaric bupivacaine is used instead of isobaric bupivacaine in continuous spinal anesthesia for surgical repair of hip fracture in elderly patients. Half of the patients will receive hypobaric bupivacaine and the over half will reveive isobaric bupivacaine and hemodynamic data will be compared.

DETAILED DESCRIPTION:
Anesthesia for surgical repair of hip fracture is still controversial. Large retrospective studies and systematic reviews failed to demonstrate the superiority of either general or regional anesthesia. However, continuous spinal anesthesia has been shown to preserve hemodynamics better than general and single shoot spinal anesthesia. However, hypotension still occurs with continuous spinal anesthesia.

Unilateral spinal anesthesia may be achieved by hypobaric bupivacaine when patients are in the lateral position. Unilateral spinal anesthesia is more effective in preserving hemodynamics by limiting the spread of the sympathetic blockade to the operated side.

Our goal is to show that the use of hypobaric rather than isobaric bupivacaine in continuous spinal anesthesia for surgical repair of hip fracture reduces incidence of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 65 years and scheduled for a surgical repair of a hip fracture.

Exclusion Criteria:

* contraindication to spinal anesthesia or peripheral nerve blocks including hemostasis anomalies, local infection, allergic reaction to local anesthetics.
* dementia.
* consent refusal.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who experienced at least one episode of hypotension during surgery (fall of more than 20% of systolic blood pressure) among the 2 groups | 2 hours

SECONDARY OUTCOMES:
Total bupivacaine consumption | 2 hours
  total dose of bupivacaine needed to perform the surgery (approximate duration of surgery : 2 hours)
The percentage of patients who experienced at least one episode of bradycardia (heart rate<50 bpm) among the 2 groups | 2 hours
vasopressor use | 2 hours
  total ephedrine injected if hypotension occurred (approximate duration of surgery : 2 hours).
fluid infusion | 2 hours
  total fluid infused intravenously at the end of surgery (approximate duration of surgery : 2 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Kassab d'Orthopédie, Manouba, La Manouba, Tunisia

REFERENCES:
- [Background] Neuman MD, Rosenbaum PR, Ludwig JM, Zubizarreta JR, Silber JH. Anesthesia technique, mortality, and length of stay after hip fracture surgery. JAMA. 2014 Jun 25;311(24):2508-17. doi: 10.1001/jama.2014.6499. PMID 25058085
- [Background] Patorno E, Neuman MD, Schneeweiss S, Mogun H, Bateman BT. Comparative safety of anesthetic type for hip fracture surgery in adults: retrospective cohort study. BMJ. 2014 Jun 27;348:g4022. doi: 10.1136/bmj.g4022. PMID 24972901
- [Result] Minville V, Fourcade O, Grousset D, Chassery C, Nguyen L, Asehnoune K, Colombani A, Goulmamine L, Samii K. Spinal anesthesia using single injection small-dose bupivacaine versus continuous catheter injection techniques for surgical repair of hip fracture in elderly patients. Anesth Analg. 2006 May;102(5):1559-63. doi: 10.1213/01.ane.0000218421.18723.cf. PMID 16632842